CLINICAL TRIAL: NCT06938035
Title: Effect of H.Pylori Infection on Growth Parameters Of Primary School-aged Children Attending Assuit University Children Hospital
Brief Title: Effect of H.Pylori Infection on Growth Parameters
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed shaban Abdelqway Gomaa, 71515,Assiut, Assiut University
Other Study IDs: H.pylori infection
Record Dates: First submitted 2024-10-02; First posted 2025-04-22 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: HELICOBACTER PYLORI INFECTIONS

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study aimed to assess the effect H.pylori infection on growth parameter Of primary school-aged children Attending Assuit university chilren hospital

DETAILED DESCRIPTION:
Undernutrition is caused by insufficient intake, malabsorption, inadequate utilization, and increased demand. There is a positive association between undernutrition and various infections. Chronic exposure to pathogens may affect nutrient absorption and increase nutrient consumption, Among many potential pathogens, chronic Helicobacter pylori (H. pylori) infection may be one cause of undernutrition. H. pylori is a gram-negative, helical, and microaerophilic bacterium, which colonizes gastric epithelial cells' surface. The mode of transmission of H. pylori is not known exactly, but the faecal-oral or oral-oral routes via water or food consumption are thought to be a very common cause. The frequency of H.pylori infection increases with age. The rate of development is higher in societies with low socioeconomic status .

The worldwide prevalence of H. pylori in children varies significantly, from 2.5% in Japan to 34.6% in Ethiopia. Gastric mucosal host factors, as well as environmental and virulence factors of the bacteria, are associated with the clinical outcome of H. pylori infection. it is closely related to chronic gastritis, dyspepsia, and chronic diarrhea. H pylori also remains an important risk factor for duodenal ulcers and duodenal and gastric erosions in children.A number of studies identified correlations of H pylori infection in children with a variety of gastrointestinal diseases including autoimmune gastritis and celiac disease. It also produces different biological effects on hormones such as ghrelin and leptin, which control both growth and appetite, causing changes in appetite and food intake, while causing changes in immunological symptoms and responses .H. pylori is a factor that causes malnutrition and growth retardation, due to malabsorption of nutrients and increased susceptibility to enteric infections, especially in developing countries .

ELIGIBILITY:
Inclusion Criteria:

1. Primary school children aged 6 to 12 years old.
2. Children who have tested positive for Helicobacter pylori.

Exclusion Criteria:

1. Children with primary malnutrition due to nutritional deficiency .
2. Children with chronic illness

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: primary school-aged children Attending Assuit university hospital Of pediatrics .
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2025-05-13 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
H.pylori infection and its effect on growth parameter | baseline
  Assess the effect of H.pylori infection on growth parameter of primary school-aged children attending Assiut university children hospital by assesing :
  1. anthropometric measurement :Weigt (kg), height(cm) ,head circumference (cm),body mass index(m2/kg)
  2. cbc
  3. serum albumin
  4. stool analysis
  5. upper endoscopy

REFERENCES:
- [Background] Zamani M, Vahedi A, Maghdouri Z, Shokri-Shirvani J. Role of food in environmental transmission of Helicobacter pylori. Caspian J Intern Med. 2017 Summer;8(3):146-152. doi: 10.22088/cjim.8.3.146. PMID 28932364
- [Background] Hooi JKY, Lai WY, Ng WK, Suen MMY, Underwood FE, Tanyingoh D, Malfertheiner P, Graham DY, Wong VWS, Wu JCY, Chan FKL, Sung JJY, Kaplan GG, Ng SC. Global Prevalence of Helicobacter pylori Infection: Systematic Review and Meta-Analysis. Gastroenterology. 2017 Aug;153(2):420-429. doi: 10.1053/j.gastro.2017.04.022. Epub 2017 Apr 27. PMID 28456631